CLINICAL TRIAL: NCT00756210
Title: Lifestyle and Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College of Antwerp (Other)
Other Study IDs: DepG0002
Record Dates: First submitted 2008-09-18; First posted 2008-09-22 (Estimated); Last update posted 2008-09-22 (Estimated); Status verified 2008-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

INTERVENTIONS:
Other: Whole body vibration — Frequence: 35 Hz Amplitude: 'high' (approx. 4 mm)

SUMMARY:
The objective of this trial is to determine the effect of different lifestyle interventions such as aerobic exercise and alternative resistance training methods, combined with a hypocaloric diet, on weight, body composition and metabolic risk factors in overweight and obese adults.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index > 24.9 kg/m²
* age > 18 y
* pre-menopauzal

Exclusion Criteria:

* Body mass index > 40 kg/m²
* Pregnancy
* Diabetes
* Joint replacement surgery

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium